| Dementia Awareness Course UK Study |
|---|
| Investigating the Feasibility, Acceptability, and Impact of an Online UK Dementia Awareness<br>Course for Informal Caregivers: A Mixed Methods Study |
| Document date: 7 <sup>th</sup> June 2022 |
| Document date. 7° June 2022 |

## CONSENT FORM

UCL Research Ethics Committee Approval ID Number: 22375/001

| <b>Title of Study:</b> Investigating the feasibility, acceptability and impact of an online UK "Dementia Awareness Course for unpaid caregivers. | <u>"'</u> ڊ |
|---|---|
| <b>Department:</b> Clinical, Educational and Health Psychology, Faculty of Brain Sciences, Division of Psychology and Language Sciences, UCL | |
| Name and Contact Details of the Researcher(s): Ria Patel (r.patel.20@ucl.ac.uk) & Izzy Evans (izzy.evans.20@ucl.ac.uk) Name and Contact Details of the Principal Researcher: Professor Aimee Spector (a.spector@ucl.ac.uk) Name and Contact Details of the UCL Data Protection Officer: This study has been approved by the UCL Research Ethics Committee: Project ID number: | |

Please complete this form after you have read the Information Sheet and/or listened to an explanation about the research.

Thank you for considering taking part in this research. The person organising the research must explain the project to you before you agree to take part. If you have any questions arising from the Information Sheet or explanation already given to you, please ask the researcher before you decide whether to join in. You will be given a copy of this Consent Form to keep and refer to at any time.

I confirm that I understand that by ticking/initialling each box below I am consenting to this element of the study. I understand that it will be assumed that unticked/initialled boxes means that I DO NOT consent to that part of the study. I understand that by not giving consent for any one element that I may be deemed ineligible for the study.

| Parti | cipant Identification Number for this project: | <br>_ |
|---|---|---|
| 1 | I confirm that I have read and understood the Participant Information Sheet | |
| | dated 02.2022 for the above project. I have had the opportunity to consider | |
| | this information, ask questions and have had these answered satisfactorily. | |
| 2 | I understand that my participation is voluntary and that I am free to withdraw | |
| | at any time without giving any reason, up until data analysis. I understand that | |
| | if I decide to withdraw, any personal data I have provided up to that point will | |
| | be deleted unless I agree otherwise. | |

| 3 | I consent to participate in the study. I understand that my personal |
|---|---|
| | information (age, ethnicity, gender, telephone number, email address) will be |
| | used for the purposes explained to me. I understand that according to data |
| | protection legislation, 'public task' will be the lawful basis for processing. |
| 4 | Use of the information for this project only |
| | I understand that all personal information will remain confidential and that all |
| | efforts will be made to ensure I cannot be identified (unless you state |
| | otherwise, because of the research design or except as required by law). |
| | I understand that my data gathered in this study will be stored anonymously |
| | and securely. It will not be possible to identify me in any publications. |
| 5 | I understand that my information may be subject to review by responsible |
| | individuals from the University (to include sponsors and funders) for |
| | monitoring and audit purposes. |
| 6 | I understand the direct/indirect benefits of participating. |
| 7 | I understand that the data will not be made available to any commercial |
| | I understand that the data will not be made available to any commercial organisations but is solely the responsibility of the researcher(s) undertaking |
| 7 | I understand that the data will not be made available to any commercial organisations but is solely the responsibility of the researcher(s) undertaking this study. |
| | I understand that the data will not be made available to any commercial organisations but is solely the responsibility of the researcher(s) undertaking |
| 7 | I understand that the data will not be made available to any commercial organisations but is solely the responsibility of the researcher(s) undertaking this study. |
| 7 | I understand that the data will not be made available to any commercial organisations but is solely the responsibility of the researcher(s) undertaking this study. I understand that I will not benefit financially from this study or from any |
| 7 8 | I understand that the data will not be made available to any commercial organisations but is solely the responsibility of the researcher(s) undertaking this study. I understand that I will not benefit financially from this study or from any possible outcome it may result in in the future. |
| 7 8 | I understand that the data will not be made available to any commercial organisations but is solely the responsibility of the researcher(s) undertaking this study. I understand that I will not benefit financially from this study or from any possible outcome it may result in in the future. If I am asked to engage in an interview as part of the study, I consent to my |
| 7 8 | I understand that the data will not be made available to any commercial organisations but is solely the responsibility of the researcher(s) undertaking this study. I understand that I will not benefit financially from this study or from any possible outcome it may result in in the future. If I am asked to engage in an interview as part of the study, I consent to my interview being audio recorded and understand that the recordings will be |
| 7 8 | I understand that the data will not be made available to any commercial organisations but is solely the responsibility of the researcher(s) undertaking this study. I understand that I will not benefit financially from this study or from any possible outcome it may result in in the future. If I am asked to engage in an interview as part of the study, I consent to my interview being audio recorded and understand that the recordings will be stored anonymously, using password-protected software and destroyed |
| 8 | I understand that the data will not be made available to any commercial organisations but is solely the responsibility of the researcher(s) undertaking this study. I understand that I will not benefit financially from this study or from any possible outcome it may result in in the future. If I am asked to engage in an interview as part of the study, I consent to my interview being audio recorded and understand that the recordings will be stored anonymously, using password-protected software and destroyed immediately following transcription. |

Dementia Awareness Course UK Study

| <br>Nam | | - |
|---|---|---|
| | | l |
| 13 | I voluntarily agree to take part in the above project. | |
| 12 | I am aware of who I should contact if I wish to lodge a complaint. | |
| 11 | I hereby confirm that I understand the inclusion criteria as detailed in the Information Sheet and explained to me by the researcher. | |
| 11 | I horaby confirm that I understand the inclusion criteria as detailed in the | |